CLINICAL TRIAL: NCT05760469
Title: Seeing Red: Towards Improving 'Recognition, Documentation and Outcome 'Measurement of Incontinence-associated 'Dermatitis and Intertrigo
Brief Title: Seeing Red: Clinical Assessment Tools for Clinical Trial Decision Support
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scotiaderm (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Seeing Red
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Incontinence-associated Dermatitis; Moisture Associated Skin Damage; Intertrigo
MeSH Terms: conditions — Intertrigo | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: Data for this study will be collected daily until you are discharged from the hospital, up to a maximum of 7 days. Study data will be collected by the nurses/research assistants during regular patient check-ins and will require minimal time to complete (15-20min maximum). Participants for the study will be identified by nursing staff from patients admitted to the Valley Regional Hospital. After informed consent, where possible, the primary care nurse will collect qualitative information from the patient based on the history of their skin condition, whether the rash is new or recurring for them, and their pain, irritation, and discomfort measures. All patients participating in the study will receive the standard of care for patients presenting with MASD as prescribed by their primary care physician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening Rash (Other): This is an exploratory study to assess the usefulness and reliability of the ITD-IAD-M for diagnosing, tracking, and treating IAD and ITD in hospitals.Participants for the study will be identified by nursing staff from admitted patients. After informed consent, the primary care nurse will collect qualitative information from the patient based on the history of their skin condition, whether the rash is new or recurring for them, and their pain, irritation, and discomfort measures. All patients participating in the study will receive the standard of care for patients presenting with MASD as prescribed by their primary care physician. The nurse will complete the ITD-IAD-M tool daily along with routine patient care. Each day the nurse documents the rash status and whether the treatment can be stopped based on the nursing assessment. The nurse/research assistant will also take a standardized digital live picture of the rash (without any identifying features) daily for a maximum of 7 days.
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Clinical nurse (CN) notifies research coordinator (RC) about patients with rashes. RC assesses eligibility criteria of patient based on inclusion criteria. RC provide CN with appropriate documentation tool (DT), smart device (SD), standardized red adhesive label (SRAL), and adhesive QRcode. Intervention: With written informed consent, demographic information will be collected. QRcode adhesive will be placed in the DT to track subject documentation throughout the study. Baseline live photograph (LP) of the rash will be taken with SD at day 0. LP will be taken daily. A SRAL, and a QR adhesive code will be included in the LP. LP will be automatically saved in a secure file on the cloud server under the QR code. CN will complete the DT for all rashes included in the study. Treatment of the rash will be at the discretion of the clinical team; the treatment regimen will be recorded daily. The procedure will be repeated daily for all rashes during the patient stay to a maximum of 7 days.

SUMMARY:
This research aims to assess the utility and validate the inter-rater reliability of the new nursing documentation tools for commonly encountered moisture-associated skin damage including (incontinence-associated dermatitis (IAD) and intertrigo (ITD)) at Valley Regional Hospital.

This is an exploratory study to assess the utility and accuracy of a structured documentation tool for IAD and ITD in hospitals. Current documentation involves a mostly verbal description of the location, size, and general features of the rash. Without a standardized approach to documentation, it can be challenging to accurately evaluate the evolution of the rash and the response to treatment from day to day and from different nurses. The reliability of the documentation tool will be assessed by comparing the results of the bedside assessment tool with that completed by wound care experts using standardized digital live photographs. The utility documentation tool from a nursing perspective will also be assessed using a structured questionnaire. Analysis of digital live photographs using a standard algorithm will be done to determine whether such an analysis can objectively and accurately track the healing of moisture-associated skin damage.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Intertrigo (ITD) and or incontinence-associated dermatitis (IAD)
* Expected length of stay of seven (7) days
* life expectancy greater than one week
* written informed consent by the patient or his/her representative including explicit consent to take daily photographs of the rash associated with MASD.

Exclusion Criteria:

* known allergy to standard MASD treatments
* life expectancy less than seven days
* complex skin disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
ITD-IAD-M Assessment tool | 7 days
  The primary outcome measurement is the correlation between the assessment of the rash by the primary care nurse and the assessment by the wound care expert, with respect to the categorization of the rash, the surface area involvement, and the timing of termination of treatment.

IPD SHARING:
Plan to Share IPD: No
The study data will not be shared with other researchers.